CLINICAL TRIAL: NCT04468321
Title: Heart Watch Study: a Pragmatic Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Mayo Clinic (Other); Duke University (Other); National Evaluation System for health Technology Coordinating Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000028126; 6292-2020-R2TC-T12T13 (Other Grant/Funding Number: Medical Device Innovation Consortium, on behalf of the NESTcc)
Record Dates: First submitted 2020-07-07; First posted 2020-07-13 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Cardioversion; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Apple Watch (Experimental): Patients will be provided with the Apple Watch Series 6 with Irregular Rhythm Detection and ECG capabilities.
  Interventions: Device: Apple Watch
- Withings Move (Placebo Comparator): Patients will be provided with the Withings Move with activity tracking.
  Interventions: Device: Withings Move

INTERVENTIONS:
Device: Apple Watch — Participants will be assigned to the Apple Watch arm to assess the impact of individual use of the Apple Watch on patient-reported and clinical utilization outcomes using Hugo.
  Arms: Apple Watch
Device: Withings Move — Participants will be assigned to the Withings Move arm to assess the impact of individual use of the Withings Move on patient-reported and clinical utilization outcomes using Hugo.
  Arms: Withings Move

SUMMARY:
This will be a prospective multi-center, randomized, controlled trial of 150 patients conducted to assess the impact of individual use of the Apple Watch compared to the Withings Move on patient-reported and clinical outcomes at 6 months and up to 1 year.

DETAILED DESCRIPTION:
This is a a randomized, controlled trial to determine the impact of the Apple Watch Series 6 compared to the Withings Move on both patient-reported outcomes and clinical utilization over 6 months and up to 1 year. Our research method will employ a patient-centered health data sharing platform (called Hugo) for real-world surveillance of outcomes in 150 total patients after they receive elective direct current cardioversion (DCCV) or catheter ablation for treatment of atrial fibrillation or atrial flutter. Patients will be enrolled at each of 3 clinical sites: Yale-New Haven Hospital, the Mayo Clinic, and Duke Health. Half of the patients will be randomized to receive the Apple Watch Series 6, while half will receive a control device (Withings Move). Patients will then be queried about specific symptoms related to atrial fibrillation and medication adherence monthly. This project will provide novel and needed post-market data about the Apple Watch Series 6 ECG and irregular rhythm detection notification features and, on a larger scale, help delineate the impact of an innovative digital health technology on real-world patient outcomes.

Specific Aim 1: To assess the impact of using the Apple Watch ECG and irregular rhythm notification features on patient-reported outcomes and clinical utilization after patients receive cardioversion or catheter ablation for atrial fibrillation or atrial flutter.

Specific Aim 2: To determine the accuracy of the Apple Watch ECG compared to physician interpretation of 12-lead ECGs obtained in routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age >22
* English-speaking
* Planned for direct current cardioversion or catheter ablation for atrial fibrillation or atrial flutter, as noted by referring clinical staff or on chart review
* Participant is willing and able to read and sign consent and participate in study
* Participant lives independently and does not require continuous care
* Participant has an email account (or is willing to create one)
* Participant has a compatible smartphone (iPhone 6s or later)
* Participant is willing to wear only the device they are randomized to receive for the study period for as many hours during the day as they are able, except for time spent charging the device or in environments that may be suboptimal for the device
* Participant is willing to use the Hugo mobile health platform and Apple Watch Series 6 or Withings Move
* Participant has cardiology care at YNHH, Duke Health, or Mayo Clinic

Exclusion Criteria:

* No exclusion criteria

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ross, MD, MHS, Principal Investigator — Yale University; Peter Noseworthy, MD, Principal Investigator — Mayo Clinic; Sreekanth Vemulapalli, MD, Principal Investigator — Duke University; Sanket Dhruva, MD, MHS, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Once the study has been completed, IPD will be shared in a way which will protect patient confidentiality using a data sharing platform for research purposes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available once the study has been completed.

REFERENCES:
- [Derived] Dhruva SS, Shah ND, Vemulapalli S, Deshmukh A, Beatty AL, Gamble GM, Freeman JV, Hummel JP, Piccini JP, Akar JG, Ervin K, Arges KL, Emanuel L, Noseworthy PA, Hu T, Bartlett V, Ross JS. Heart Watch Study: protocol for a pragmatic randomised controlled trial. BMJ Open. 2021 Dec 30;11(12):e054550. doi: 10.1136/bmjopen-2021-054550. PMID 35234659
- See also: Preprint of protocol manuscript — https://medrxiv.org/cgi/content/short/2021.07.10.21260230v1

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apple Watch | Withings Move
Started | 70 | 35
Completed | 60 | 25
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apple Watch | Withings Move | Total
Number analyzed (Participants) | 70 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.22) | 70.3 (9.55) | 66.9 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 51 | 25 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska Native | 1 | 0 | 1
  Race/Ethnicity: Black or African American | 2 | 3 | 5
  Race/Ethnicity: Black or African American and White | 0 | 1 | 1
  Race/Ethnicity: White | 67 | 31 | 98

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life)
Description: Change in the Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) questionnaire global score at 6 months compared to baseline between the Apple Watch and patients randomized to the Withings Move arm at 6 months compared to baseline. Reported on a scale from 0 to 100 with a higher score indicating a better outcome.
Time Frame: baseline and 6 months
Population: Number of patients that completed the AFEQT questionnaire at 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 60 | 25
score on a scale | 20.3 [14.7 to 25.8] | 17.9 [8.6 to 27.2]

2. Secondary Outcome: Change in Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life)
Description: Change in the Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) questionnaire global score at 12 months compared to baseline between the Apple Watch and patients randomized to the Withings Move arm at 12 months compared to baseline. Reported on a scale from 0 to 100 with a higher score indicating a better outcome.
Time Frame: baseline and 12 months
Population: Number of patients that completed the AFEQT questionnaire at 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 43 | 12
score on a scale | 23.5 [16.6 to 30.4] | 25.0 [11.0 to 39.1]

3. Secondary Outcome: Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life) Domain- Symptoms
Description: Difference within individual Symptoms domain of the Atrial Fibrillation Effect on QualiTy-of-life questionnaire between patients randomized to the Apple Watch and patients randomized to the Withings Move arm over the 6-month period. Reported on a scale from 0 to 100 with a higher score indicating a better outcome
Time Frame: 6 months
Population: Number of patients that completed the AFEQT Questionnaire at 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 60 | 25
score on a scale | 21.8 [14.0 to 29.5] | 13.1 [6.0 to 20.2]

4. Secondary Outcome: Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life) Domain- Symptoms
Description: Difference within individual Symptom domain of the Atrial Fibrillation Effect on QualiTy-of-life questionnaire between patients randomized to the Apple Watch and patients randomized to the Withings Move arm over the 12-month period. Reported on a scale from 0 to 100 with a higher score indicating a better outcome
Time Frame: 12 months
Population: Number of patients that completed the AFEQT questionnaire at 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 43 | 12
score on a scale | 23.7 [15.8 to 31.6] | 25.3 [10.5 to 40.1]

5. Secondary Outcome: Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life) Domain- Daily Activities
Description: Difference within individual Daily Activities domain of the Atrial Fibrillation Effect on QualiTy-of-life questionnaire between patients randomized to the Apple Watch and patients randomized to the Withings Move arm over the 6-month period. Reported on a scale from 0 to 100 with a higher score indicating a better outcome
Time Frame: 6 months
Population: Number of patients that completed the AFEQT Questionnaire at 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 60 | 24
score on a scale | 22.1 [14.7 to 29.5] | 20.5 [8.6 to 32.4]

6. Secondary Outcome: Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life) Domain- Daily Activities
Description: Difference within individual Daily Activities domain of the Atrial Fibrillation Effect on QualiTy-of-life questionnaire between patients randomized to the Apple Watch and patients randomized to the Withings Move arm over the 12-month period. Reported on a scale from 0 to 100 with a higher score indicating a better outcome
Time Frame: 12 months
Population: Number of patients that completed the AFEQT questionnaire at 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 42 | 12
score on a scale | 27.2 [18.4 to 36.0] | 27.2 [8.2 to 46.2]

7. Secondary Outcome: Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life) Domain- Treatment Concern
Description: Difference within individual Treatment Concern domain of the Atrial Fibrillation Effect on QualiTy-of-life questionnaire between patients randomized to the Apple Watch and patients randomized to the Withings Move arm over the 6-month period. Reported on a scale from 0 to 100 with a higher score indicating a better outcome
Time Frame: 6 months
Population: Number of patients that completed the AFEQT Questionnaire at 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 60 | 24
score on a scale | 17.1 [11.4 to 22.7] | 21.0 [10.5 to 31.5]

8. Secondary Outcome: Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life) Domain- Treatment Concern
Description: Difference within individual Treatment Concern domain of the Atrial Fibrillation Effect on QualiTy-of-life questionnaire between patients randomized to the Apple Watch and patients randomized to the Withings Move arm over the 12-month period. Reported on a scale from 0 to 100 with a higher score indicating a better outcome
Time Frame: 12 months
Population: Number of patients that completed the AFEQT questionnaire at 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 43 | 12
score on a scale | 17.6 [10.0 to 25.2] | 21.9 [8.6 to 35.3]

9. Secondary Outcome: Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life) Domain- Treatment Satisfaction
Description: Difference within individual Treatment Satisfaction domain of the Atrial Fibrillation Effect on QualiTy-of-life questionnaire between patients randomized to the Apple Watch and patients randomized to the Withings Move arm over the 6-month period. Reported on a scale from 0 to 100 with a higher score indicating a better outcome
Time Frame: 6 months
Population: Number of patients that completed the AFEQT Questionnaire at 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 59 | 24
score on a scale | 19.3 [12.0 to 26.6] | 11.1 [-5.2 to 27.4]

10. Secondary Outcome: Quality-of-life (Atrial Fibrillation Effect on QualiTy-of-life) Domain- Treatment Satisfaction
Description: Difference within individual Treatment Satisfaction domain of the Atrial Fibrillation Effect on QualiTy-of-life questionnaire between patients randomized to the Apple Watch and patients randomized to the Withings Move arm over the 12-month period. Reported on a scale from 0 to 100 with a higher score indicating a better outcome
Time Frame: 12 months
Population: Number of patients that completed the AFEQT questionnaire at 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 42 | 12
score on a scale | 25.5 [16.9 to 34.2] | 25.0 [2.3 to 47.6]

11. Secondary Outcome: Proportion of Patients Taking Anticoagulants
Description: Anticoagulation use will be assessed at 6 months using the Brief Medication Questionnaire to trend patients' monthly responses about anticoagulation use
Time Frame: 6 months
Population: Responses were received for n=84 participants. Data were missing for n=21 participants.
Measure: Number; unit: percentage of patients
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 60 | 24
percentage of patients | 98.3 | 91.6

12. Secondary Outcome: Proportion of Patients Taking Anticoagulants
Description: Anticoagulation use will be assessed at 12 months using the Brief Medication Questionnaire to trend patients' monthly responses about anticoagulation use
Time Frame: 12 months
Population: Responses were received for n=55 participants. Data were missing for n=50 participants.
Measure: Number; unit: percentage of patients
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 43 | 12
percentage of patients | 90.6 | 91.6

13. Secondary Outcome: Proportion of Participants With Acute Care Use at 6 Months
Description: Acute care use will be compared between the two groups at 6 months. Acute care is defined as an emergency department visits, observation stays, and all hospitalizations over the 6 month period.
Time Frame: 6 months
Population: The emergency department visits, observation stays, and all hospitalizations data were not collected due to broken connections between the data aggregating platform and the participant's electronic health record. The team did not discover this until after the participant follow-up period concluded.
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Proportion of Participants With Acute Care Use at 12 Months
Description: Acute care use will be compared between the two groups at 12 months. Acute care is defined as an emergency department visits, observation stays, and all hospitalizations over the 12 month period.
Time Frame: 12 months
Population: as for outcome 13
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Proportion of Participants With Outpatient Care Use at 6 Months
Description: Outpatient care use will be compared between the two groups at 6 months. Outpatient care is defined as outpatient primary care visits, outpatient cardiology or cardiac electrophysiology visits, and scheduled telephone encounters.
Time Frame: 6 months
Population: The outpatient primary care visits, outpatient cardiology or cardiac electrophysiology visits, and scheduled telephone encounters data were not collected due to broken connections between the data aggregating platform and the participant's electronic health record. The team did not discover this until after the participant follow-up period concluded.
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Proportion of Participants With Outpatient Care Use at 12 Months
Description: Outpatient care use will be compared between the two groups at 12 months. Outpatient care is defined as outpatient primary care visits, outpatient cardiology or cardiac electrophysiology visits, and scheduled telephone encounters.
Time Frame: 12 months
Population: as for outcome 15
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Proportion of Participants With Rhythm-related Diagnostic Testing at 6 Months
Description: Rhythm-related diagnostic testing will be assessed at 6 month including total ECGs and total outpatient heart rhythm monitors
Time Frame: 6 months
Population: The total ECGs and total outpatient heart rhythm monitors data were not collected due to broken connections between the data aggregating platform and the participant's electronic health record. The team did not discover this until after the participant follow-up period concluded.
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Proportion of Participants With Rhythm-related Diagnostic Testing at 12 Months
Description: Rhythm-related diagnostic testing will be assessed at 12 month including total ECGs and total outpatient heart rhythm monitors
Time Frame: 12 months
Population: as for outcome 17
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Proportion of Participants With Clinical Treatment for Atrial Fibrillation or Flutter
Description: A composite outcome of rhythm control intervention, which is defined as at least one additional cardioversion, initiation of antiarrhythmic medical therapy, dose escalation of antiarrhythmic medication, change to another antiarrhythmic medication, or ablation for atrial fibrillation over the 6 month period. The medication data will be obtained primarily from electronic health record data.
Time Frame: 6 months
Population: The medication data were not collected due to broken connections between the data aggregating platform and the participant's electronic health record. The team did not discover this until after the participant follow-up period concluded.
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Proportion of Participants With Clinical Treatment for Atrial Fibrillation or Flutter
Description: A composite outcome of rhythm control intervention, which is defined as at least one additional cardioversion, initiation of antiarrhythmic medical therapy, dose escalation of antiarrhythmic medication, change to another antiarrhythmic medication, or ablation for atrial fibrillation over the 12 month period. The medication data will be obtained primarily from electronic health record data.
Time Frame: 12 months
Population: as for outcome 19
Arm/Group | Apple Watch | Withings Move
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 12 months.
Arm/Group | Apple Watch | Withings Move
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/35
Other Adverse Events (participants affected / at risk) | 0/70 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT04468321/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04468321/SAP_001.pdf
  • Informed Consent Form (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT04468321/ICF_002.pdf